CLINICAL TRIAL: NCT02739152
Title: TRIAGE: TRIage of Sepsis At emerGency dEpartment
Acronym: TRIAGE
Status: Completed | Type: Observational
Sponsor: BioMérieux (Industry)
Collaborators: Centre Investigation Clinique, Limoges (Unknown)
Responsible Party: Sponsor
Other Study IDs: TRIAGE
Record Dates: First submitted 2016-03-22; First posted 2016-04-15 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Sepsis; Severe Sepsis
Keywords: Sepsis; Severe sepsis; Infections; Worsening
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sepsis is a serious systemic disease defined as a combination of Systemic Inflammation Response Syndrome (SIRS) plus a confirmed or suspected infection. Untreated or inadequately treated cases can lead to severe sepsis or septic shock; being characterized by high mortality and morbidity.

Symptoms and signs of sepsis are variable and this makes clinical recognition and assessment very difficult in particular on Emergency Department (ED) patients due to their infectious illness background and the frequent comorbidities. Also, the severity of the condition may not be apparent at initial contact with ED personnel: patients may arrive at ED with mild clinical manifestation and rapidly progress to critical illness, or rather at the opposite others have benign evolution despite a similar symptoms. In these conditions, the main challenge of ED clinicians is differentiating mild infections from life-threatening ones in the heavy workload of ED environment Objective of TRIAGE project is to identify and validate biomarkers able to predict the clinical worsening of patients freshly admitted at Emergency Department.

Targeted population is adult patients freshly admitted at ED, whom blood samples will serve to validate candidate markers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged over 18 years
* Patient with a single acute infection site suspected or confirmed by the clinician on clinical or paraclinical manifestations.
* Patient admitted to ED with at least two systemic inflammatory response syndrome (SIRS) criteria
* Patient with symptoms for less than 72 hours upon arrival to the emergency department.
* Patient requiring according to physician judgment of hospitalization for at least 48 hours for his septic episode
* Patient having been informed of the conditions of the study and having signed the informed consent form

Exclusion Criteria:

* Patient arrived in an emergency room for over 6 hours.
* Patient with septic shock upon arrival to the ED Patient with acute organ failure on arrival at emergencies other than septic.
* Patient hospitalized in the week before inclusion.
* Patient immunocompromised (HIV, transplanted, patients undergoing chemotherapy, patients receiving treatment> 20 mg / day of prednisolone or equivalent).
* Patient with known pathology among non-infectious pathologies potentially associated with SIRS
* Patient diagnosed with sepsis within 30 days before the date of inclusion.
* Patient has already been included in the study.
* Minor Person.
* Person refusing to sign the written consent form.
* Pregnant woman parturient or nursing.
* Patient with no social security insurance, with restricted liberty or under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient freshly admitted to Emergency department
Sampling Method: Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2015-04; Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
patient worsening within a time frame of 72h,change, from day of inclusion, in Sequential Organ Failure Assessment score (SOFA) and/or sepsis classification | Up to 72 hours after admission
  A biostatistics analysis will be led in two steps. The first analysis or "train set" will be conducted on the first 150 patients enrolled, estimated size to reach statistical performance. The objective is to identify markers associated with clinical worsening of patients and decide on a model by selecting the best combination of markers. In a second time, performance will be confirmed during the "test set". The number of samples to be tested depends on the target performance calculated with the area under the Receiver operating characteristic (ROC) curve (AUC). We decided to aim for an AUC of 0.75, based on the performance described in the literature for some triage score as MEDS (Mortality in Emergency Department Sepsis) or those associated with Lactate concentration used as marker of sepsis deterioration in ED

SECONDARY OUTCOMES:
patient status at D28 (alive or death) | Up to 28 days after admission
  A biostatistics analysis will be led in two steps. The first analysis or "train set" will be conducted on the first 150 patients enrolled. The objective is to identify markers associated with mortality at day 28. In a second time, the performance will be confirmed during the "test set".

CONTACTS AND LOCATIONS:
Locations (14):
- Cliniques universitaires Saint-Luc - UCL, Brussels, Belgium
- France (13):
  - Centre hospitalier universitaire Grenoble Alpes, Grenoble, La Tronche
  - Centre Hospitalier Angoulême, Angoulême
  - Centre Hospitalier Henri Mondor, Aurillac
  - Centre Hospitalier Regional Universitaire de Besançon, Besançon
  - Centre Hospitalier Brive La Gaillarde, Brive-la-Gaillarde
  - Centre Hospitalier Départemental - Hôpital La Roche-sur-Yon, La Roche-sur-Yon
  - Centre d'Investigation Clinique (CIC)-CHU Limoges, Limoges
  - Centre Hospitalier Universitaire Edouard Herriot, Lyon
  - Centre Hospitalier de Montauban, Montauban
  - CHU Montpellier, Montpellier
  - Assistance publique - Hôpitaux de Paris Hopital de Cochin, Paris
  - Centre Hospitalier Régional Universitaire de Tours, Tours
  - Centre Hospitalier de Versailles, Versailles

IPD SHARING:
Plan to Share IPD: Yes